CLINICAL TRIAL: NCT04244240
Title: Cognitive Functions in Adults With Sickle Cell Disease and Cognitive Complaints: Neuropsychological Assessment and Links to Demographic, Clinical, Biological, Neuroradiological Outcomes and Validation of a Cognitive Assessment Tool.
Brief Title: Links Between Cognitive Functions and Clinical, Biological and Neuroradiological Outcomes in Adults With Sickle Cell Disease.
Acronym: Drépa-COG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0753; 2019-A02709-48 (Other: ID-RCB)
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Drepanocytosis
Keywords: Sickle Cell Disease; Drepanocytosis
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sickle cell disease patient: Adults with sickle cell disease (homozygous SS or heterozygous SC, Sβ0 or Sβ+) with cognitive complaint.
  Interventions: Behavioral: BEARNI Tool

INTERVENTIONS:
Behavioral: BEARNI Tool — BEARNI is brief screening tool initially validated for Alcohol-related neuropsychological impairments (Ritz et al., 2015). BEARNI tool detect impairment in visuospatial abilities, executive functions, verbal episodic memory, and verbal working memory.
  The score of the test could be expressed as a global score, and also as subscores corresponding to each cognitive subtest. Normative data are available.

SUMMARY:
Sickle cell disease (SCD) is an inherited blood disorder. Symptoms include acute and chronic complications. Due to progress in SCD care, patients with SCD are living longer than before and we focus more attention in chronic complications.

Children with SCD experience worse cognitive functions than healthy children, and fewer is known about cognitive functions in adults. Studies suggest lower cognitive performance in SCD, mostly in executive functions and processing speed, but the biological and anatomical substrates of cognitive decline are not yet well established in SCD. Often times, cognitive impairments and cerebral disorders are not diagnosed and treated in adults with SCD.

The main objective of this study is to propose a deep neuropsychological assessment in adults with SCD and cognitive complaints and to highlight links between cognitive functions and clinical, biological and neuroradiological markers. The hypothesis of this study is that cognitive functions are associated with severity of the SCD, with bood abnormalities, with MRI markers and Transcranial Doppler (TCD) markers of cerebrovascular disease. The secondary objective of this study is to validate a brief cognitive assessment tool (BEARNI tool) in adults with SCD.

This study is an observational cross-sectional study that will enroll adults with SCD and cognitive complaint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Sickle cell anemia (homozygous SS or heterozygous SC, Sβ0, S/C, Sβ+)
* In steady state (without vaso-occlusive crisis or acute chest syndrome at the time of measurements)
* Presence of spontaneous cognitive complaint or requested by the physician.
* Good command of the French language (native language or not)
* No objection to participate in the study
* Affiliated patient or beneficiary of social security scheme

Exclusion Criteria:

* Patient not compliant in the management of his disease
* Patient participating in another interventional research protocol that may interfere with this protocol (according to investigator's judgment)
* Language barrier
* Pregnancy or breast feeding
* MRI contraindication
* Patient under guardianship , curatorship or justice
* Inability to express non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sickle cell disease and cognitive complaint
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
BEARNI questionnaire | Day 0
  Cognitive performance will be evaluated by a large neuropsychological assessment. The cognitive score will be interpreted as raw scores, z-score adjusted for level of education, age, and sex, according to the tests and binarized into two categories (normal versus pathological performances)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Bron, France

IPD SHARING:
Plan to Share IPD: No